CLINICAL TRIAL: NCT05620316
Title: Evaluation of the Efficacy of Low-Dose Botulinum Toxin Injection Into the Masseter Muscle for the Treatment of Nocturnal Bruxism: A Randomized Controlled Clinical Trial
Brief Title: The Use of Low-Dose Botulinum Toxin Injection Into the Masseter Muscle to Treat Sleep Bruxism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-OMFS-02-2022
Record Dates: First submitted 2022-11-05; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Nocturnal Bruxism
Keywords: Nocturnal bruxism; Botulinum toxin; Masseter muscle; Electromyography
MeSH Terms: conditions — Sleep Bruxism | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injection group (Experimental): In this group, patients will be injected with 10 MU of botulinum toxin type A in the masseter muscle.
  Interventions: Drug: BOTOX® Injection
- Placebo group (Placebo Comparator): In this group, patients will prick twice in the masseter muscle.
  Interventions: Other: Prick skin

INTERVENTIONS:
Drug: BOTOX® Injection — 100 MU of botulinum toxin type A (BOTOX® - Allergan Inc. - Dublin - Ireland) were diluted in 2ml of saline. Patients were injected with 10 MU of BTXA per side at two sites into the masseter muscle bilaterally. The first site was the inferior prominent part of the masseter muscle observed when the subject was asked to clench, and the other site was 5 mm below the first point
  Arms: Injection group
Other: Prick skin — patients were pricked twice at the inferior prominent part of the masseter muscle observed using the stinger pen used in the blood glucose meter; it is less painful and provides psychological benefits, instead of injecting the physiological saline into the muscle to avoid the severe pain without a benefit to the patient which would not conform to the ethical standards.
  Arms: Placebo group

SUMMARY:
Botulinum toxin (BOTOX®) injections into the masseter muscle are an effective treatment for nocturnal bruxism, with several trials using various dosages of botulinum toxin for this purpose. The aim was to evaluate the effectiveness of injecting 10MU of botulinum toxin A (BTXA) into the masseter muscle to reduce nocturnal bruxism, the sample will randomly divided into 2 groups.

In the injection group, Patients will inject with 10 MU of botulinum toxin type A (BOTOX® - Allergan Inc. - Dublin - Ireland) per side at two sites into the masseter muscle bilaterally.

In this Placebo group, patients will prick twice at the inferior prominent part of the masseter muscle observed using the stinger pen used in the blood glucose meter.

The evaluation will make by Electromyography (EMG) analysis, Visual Analogue Scale (VAS) values.

DETAILED DESCRIPTION:
Nocturnal bruxism (NB) is a disorder of maxillomandibular activity characterized by nonfunctional grinding and clenching of teeth while sleeping.

NB can cause teeth attrition, dental prostheses/implant failure, tooth sensitivity, pain in the teeth, jaw, masticatory muscle, and temporomandibular joint (TMJ), neck pains and headache, periodontal disease, oral or facial pain, and perhaps tooth loss. The diagnosis of nocturnal bruxism is based on complaints of tooth grinding or clenching, as well as one or more of the following signs: nonfunctional teeth attrition, sounds consistent with bruxism, and jaw muscle discomfort. Teeth wear and TMJ dysfunction can both be caused by bruxism. In some circumstances, delaying therapy might lead to luxation and degenerative arthritis of the temporomandibular joint.

For the treatment of bruxism, many treatment approaches such as occlusal splints and pharmacologic medications such as psychobehavioral therapy or L-dopa, and psychobehavioral therapy have been examined but is not enough evidence to define a standard of reference approach for SB treatment.

Botulinum toxin (Botox®) is an exotoxin generated by the bacteria Clostridium botulinum that causes muscle inactivity by blocking acetylcholine release from cholinergic nerve terminals into the neuromuscular junction. In the last two decades, several studies have been conducted to investigate the efficacy of botulinum toxin type A (BTXA) in reducing nocturnal bruxism, and the results have been promising. These studies have used different doses of botulinum toxin ranging from 20 mouse units (MU) and 25 MU to 30 MU in the masseter. Most of these studies did not take into account the relationship between the amount of botulinum toxin dose and alteration of the masseter muscle's size and the shape of the lower third of the face, where injection of more than 20 MU into the masseter muscle affects its size and is an effective treatment for masseter muscle hypertrophy for at least 9 months. To avoid the unwanted side effects of doses greater than 20 MU, the trial aimed to evaluate the effectiveness of injecting 10 MU of the Botulinum toxin into the masseter muscle in reducing the nocturnal bruxism.

The idea of the research will explain to all patients, and the information sheets will distribute to them, then their consent will obtain.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate to severe pain in the masseter muscles during clinical examination.
2. Age range between 18 and 40 years.
3. Tooth-grinding sounds corroborated by family members or caregivers.
4. Attrition in occlusal surface of posterior teeth.

Exclusion Criteria:

1. Loss two posterior teeth or more (except for third molars).
2. Fixed or movable prosthodontics for more than four dental units.
3. Advanced malocclusion (Class II occlusion Model II - deep bite - open bite).
4. Temporomandibular disorders.
5. Pain in the orofacial region.
6. Insomnia.
7. Known botulinum toxin allergy.
8. Pregnancy.
9. Neuromuscular disease.
10. Bleeding disorders.
11. Antibiotic therapy, pulmonary disease that produced coughing during sleep.
12. Infectious skin lesion at the site of the injection.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Change in the electromyographic recorded values | Assessment will be done before the injection (T0) and then at 2 weeks (T1), 3 months (T2), and 6 months after the injection (T3)
  EMG signals will record with Matrix EP Light EMG (Micromed, Via Giotto, Mogliano Veneto, Italy) with four channels. The recorded signals will amplify sampled at 1024 Hz, and the acquired data will analyze with System Plus Evaluation software (Micromed, Via Giotto, Mogliano Veneto, Italy).
  The acquisitions will perform twice with the rest position of the mandible (RPM) for 10 seconds, in maximal intercuspal position (MIP) for five seconds and maximal teeth clenching (MTC) with 10-mm thick cotton rolls between the posterior teeth for five seconds, bilaterally, and the values obtained will be averaged.
Change in the perception of pain | Assessment will be done before the injection (T0) and then at 2 weeks (T1), 3 months (T2), and 6 months after the injection (T3)
  A visual analog scale (VAS) will be used for this assessment. A line of 100 mm in length will be used, and the patient will ask to put a mark on the line that reflects her/his perceived pain; the scores of the scale will be determined by measuring the distance in mm from the beginning to the point indicated by the patient (point (0): no pain and point (100): the highest levels of pain).

SECONDARY OUTCOMES:
Time to first observation of positive effects | 2 week
  The mean time that the effects were first seen will be recorded.
Loss of effectiveness and side effects | 4 month
  The mean time at which the loss of effectiveness started seen will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Zaed Ghassan Shehri, DDS, Principal Investigator — Department of Maxillofacial and oral surgery, Damascus University, Syria.; Issam Alkhouri, DDS,MSc,PhD, Study Director — Department of Maxillofacial and oral surgery, Damascus University, Syria.; Ibrahim Haddad, MSc,PhD, Study Director — Department of Basic Sciences, Damascus University, Syria
Locations (1):
- University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manfredini D, Ahlberg J, Winocur E, Lobbezoo F. Management of sleep bruxism in adults: a qualitative systematic literature review. J Oral Rehabil. 2015 Nov;42(11):862-74. doi: 10.1111/joor.12322. Epub 2015 Jun 11. PMID 26095208
- [Background] Carra MC, Huynh N, Lavigne G. Sleep bruxism: a comprehensive overview for the dental clinician interested in sleep medicine. Dent Clin North Am. 2012 Apr;56(2):387-413. doi: 10.1016/j.cden.2012.01.003. PMID 22480810
- [Background] Lavigne GJ, Khoury S, Abe S, Yamaguchi T, Raphael K. Bruxism physiology and pathology: an overview for clinicians. J Oral Rehabil. 2008 Jul;35(7):476-94. doi: 10.1111/j.1365-2842.2008.01881.x. PMID 18557915
- [Background] Lobbezoo F, Ahlberg J, Glaros AG, Kato T, Koyano K, Lavigne GJ, de Leeuw R, Manfredini D, Svensson P, Winocur E. Bruxism defined and graded: an international consensus. J Oral Rehabil. 2013 Jan;40(1):2-4. doi: 10.1111/joor.12011. Epub 2012 Nov 4. PMID 23121262
- [Background] Sellin LC, Thesleff S. Pre- and post-synaptic actions of botulinum toxin at the rat neuromuscular junction. J Physiol. 1981 Aug;317:487-95. doi: 10.1113/jphysiol.1981.sp013838. PMID 6273549
- [Background] Tan EK, Jankovic J. Treating severe bruxism with botulinum toxin. J Am Dent Assoc. 2000 Feb;131(2):211-6. doi: 10.14219/jada.archive.2000.0149. PMID 10680389